CLINICAL TRIAL: NCT06005480
Title: Understanding Rebound Pain After Regional Anesthesia Resolution: Mechanistic Trial in Healthy Volunteers
Brief Title: Understanding Rebound Pain After Regional Anesthesia Resolution in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Yun-Yun K. Chen, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2023P001767
Record Dates: First submitted 2023-07-16; First posted 2023-08-22 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2024-06

CONDITIONS: Regional Anesthesia Morbidity; Pain, Acute; Healthy
Keywords: Healthy volunteer; Regional anesthesia; Rebound pain
MeSH Terms: conditions — Acute Pain | interventions — Mepivacaine; Prilocaine

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to which arm will receive a nerve block.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Block upper extremity (arm) (Experimental): Upper extremity with a nerve block
  Interventions: Drug: Mepivacaine
- Control upper extremity (arm) (No Intervention): Upper extremity without a nerve block

INTERVENTIONS:
Drug: Mepivacaine — Injection of 1.5% Mepivacaine in nerve block
  Other Names: Prilocaine
  Arms: Block upper extremity (arm)

SUMMARY:
Regional anesthesia decreases postoperative pain scores and opioid consumption, and may prevent chronic pain after surgery in patients undergoing surgery. However, some patients experience an increase of pain into the severe range when the nerve block wears off, also known as rebound pain. The investigators are studying if a nerve block (numbing injection) in the arm causes hyperalgesia (increased pain) when the nerve block is wearing off.

DETAILED DESCRIPTION:
This is a prospective, randomized study in healthy volunteers who will undergo sensory testing using quantitative sensory testing (QST), complete psychosocial and pain questionnaires, and ultrasound-guided peripheral nerve block of the arm (axillary nerve block) in a supervised, monitored setting (BWH Clinical Investigation Center). The investigators plan to assess the association between different QST modalities at different time points pre- and post-nerve block resolution. Semi-structured interviews and qualitative analysis will be used to explore patient's experiences with nerve block placement.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old, ≤ 65 years old
* BMI >18, < 35
* Able to speak and understand English
* Willingness to undergo psychophysical testing (e.g., QST, pain questionnaires)
* Willingness to have nerve block performed

Exclusion Criteria:

* Ongoing acute or chronic pain in upper extremities
* Skin or tissue infection affecting upper extremities
* Previous hypersensitivity to mepivacaine or lidocaine
* Previous neuropathy (numbness, paresthesia, or motor weakness) in either upper extremity
* Loss of any limb
* Bleeding issues or bleeding disorder
* History of alcohol or drug abuse
* Currently pregnant or breastfeeding
* History of seizure or epilepsy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-09-28 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-05-28 (Actual)

PRIMARY OUTCOMES:
Heat pain detection threshold at time 1 hr | 1 hour after nerve block resolution
  Heat pain detection threshold (°C) between block arm and control arm using a heat probe at 1 hour after nerve block resolution

SECONDARY OUTCOMES:
Heat pain detection threshold and tolerance | 0-3 hours after nerve block resolution
  Heat pain detection threshold and tolerance (°C) between block arm and control arm using a heat probe at different time points up to 3 hours nerve block resolution
Pressure pain threshold and tolerance | 0-3 hours after nerve block resolution
  Pressure pain threshold and tolerance (N of force) between block arm and control arm using an algometer at different time points up to 3 hours nerve block resolution
Temporal summation and sharp pain | 0-3 hours after nerve block resolution
  Temporal summation and sharp pain (evaluated by numerical rating scale 0-10 pain score) between block arm and control arm using a pinprick device at different time points up to 3 hours nerve block
Light touch detection | 0-3 hours after nerve block resolution
  Light touch detection (mN of force) between block arm and control arm using von Frey filaments at different time points up to 3 hours nerve block
Light touch pain threshold | 0-3 hours after nerve block resolution
  Light touch pain threshold (mN of force) between block arm and control arm using von Frey filaments at different time points up to 3 hours nerve block

OTHER OUTCOMES:
Temperature change | 6-8 hours
  To observe the change in temperature between block arm and control arm (°C) pre, during, and post nerve block
Patient's experiences with nerve block | 6-8 hours
  Semi-structured interviews will be used to explore patient's experiences with nerve block placement using an immersion/crystallization approach to identify emergent themes
Pain catastrophizing and gender differences | 6-8 hours
  Correlation between situational pain catastrophizing (0-24 scale) and gender

CONTACTS AND LOCATIONS:
Overall Officials: Yun-Yun K Chen, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mass General Brigham Rally Flyer — https://rally.massgeneralbrigham.org/study/rebound_pain_nerve_block